CLINICAL TRIAL: NCT03023592
Title: A Preliminary Efficacy Study of Iguratimod in Patients With Sjögren's Syndrome
Brief Title: Study of Iguratimod in Sjögren's Syndrome
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PUMCH170115
Record Dates: First submitted 2017-01-15; First posted 2017-01-18 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Sjogren's Syndrome
Keywords: Sjogren's Syndrome; Iguratimod
MeSH Terms: conditions — Sjogren's Syndrome | interventions — iguratimod; T 614

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Iguratimod (Experimental): Patients are treated with Iguratimod 25 mg Twice a day for 24 weeks.
  Interventions: Drug: Iguratimod

INTERVENTIONS:
Drug: Iguratimod — Iguratimod 25 mg orally twice a day for 24 weeks
  Other Names: T-614

SUMMARY:
A single-center, self-control, open-label study of efficacy and safety of Iguratimod in patients with Sjögren's Syndrome

DETAILED DESCRIPTION:
In this study, patients with Sjögren's Syndrome are enrolled and received Iguratimod 25 mg twice a day for 24 weeks. The differences of ESSPRI (EULAR Sjogren's Syndrome Patient Reported Index) score, ESSPRI(EULAR Sjogren's Syndrome Patient Reported Index) score, unstimulated salivary flow rate, Schirmer's test SF-36 score and HAQ score between baseline and week 24 are evaluated to determine the efficacy of Iguratimod in patients with Sjögren's Syndrome.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of Sjogren's syndrome according to the revised American-European Consensus Group (AECG) criteria
* Positive dry eyes and (or) dry mouth symptoms
* Hyperglobulinemia

Exclusion Criteria:

* Complicated with other systemic autoimmune diseases
* Severe complications of Sjogren's syndrome
* Glucocorticosteroid therapy, systemic immunosuppressant therapy, or biological agents therapy within 3 months prior to the screening visit
* Active infections or chronic infectious diseases
* A history of malignancies
* Pregnancy or breathfeeding
* Inability to comply with the study protocol for any other reason

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-02; Primary Completion 2018-02 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
ESSDAI improvement | week 24
  The change from baseline in ESSDAI (EULAR Sjogren's Syndrome Disease Activity Index) score at 24 weeks.
ESSPRI improvement | week 24
  The change from baseline in ESSPRI (EULAR Sjogren's Syndrome Patient Reported Index) score at 24 weeks.

SECONDARY OUTCOMES:
Unstimulated salivary flow rate | week 24
  The change from baseline in unstimulated salivary flow rate at 24 weeks.
Schimer's test | week 24
  The change from baseline in Schimer's test at 24 weeks.
SF-36 | week 24
  The change from baseline in SF-36 score at 24 weeks.
HAQ | week 24
  The change from baseline in HAQ score at 24 weeks.
Immunoglobulins | week 24
  The change from baseline in IgG, IgM and IgA levels at 24 weeks.
Rheumatoid Factors | week 24
  The change from baseline in titer of rheumatoid factors at 24 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Yan Zhao, Dr., Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No